CLINICAL TRIAL: NCT06741423
Title: Distinguishing Retroperitoneal Fibrosis and Sarcoma from Other Retroperitoneal Diseases on CT Scans Via an Extended-Radiomics Approach: a Multi-Centric, International Retrospective Analysis.
Brief Title: Distinguishing Retroperitoneal Fibrosis and Sarcoma from Other Retroperitoneal Diseases Via Radiomics
Status: Active, not recruiting | Type: Observational
Sponsor: Heidelberg University (Other)
Responsible Party: Principal Investigator, Cui Yang, Private Lecturer Dr. med., Heidelberg University
Other Study IDs: 2023-890-AF 11
Record Dates: First submitted 2024-06-24; First posted 2024-12-19 (Actual); Last update posted 2024-12-19 (Actual); Status verified 2024-12

CONDITIONS: Retroperitoneal Sarcoma; Retroperitoneal Fibrosis
Keywords: radiomics; auto-segmentation
MeSH Terms: conditions — Retroperitoneal Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- retroperitoneal fibrosis: All recruited patients with retroperitoneal fibrosis
  Interventions: Other: Radiomics Algortihm
- retroperitoneal sarcoma: All recruited patients with retroperitoneal sarcoma
  Interventions: Other: Radiomics Algortihm
- other retroperitoneal diseases: All recruited patients with other retroperitoneal malignancies
  Interventions: Other: Radiomics Algortihm

INTERVENTIONS:
Other: Radiomics Algortihm — A radiomics algorithm designed to distinguish retroperitoneal fibrosis from other retroperitoneal tumors and provide recommendations for clinical treatment decisions.

SUMMARY:
A retrospective study utilizing archived CT scans of patients diagnosed with retroperitoneal fibrosis, sarcoma or other malignancies (i.e. lymphoma, germ cell tumors, metastasis, infections, ganglioneuromas) in order to implement a radiomics algorithm which is able to differentiate between these malignancies.

DETAILED DESCRIPTION:
The aim of this project is to develop a radiomics algorithm that can reliably identify retroperitoneal fibrosis (Ormond's disease) and retroperitoneal sarcomas, automatically segment them and differentiate them from other retroperitoneal diseases. Radiomics is a technique that uses artificial intelligence to extract characteristics from radiological image data that are not visible to humans and to identify image morphological patterns of diseases. As it is difficult to differentiate between diseases using image data alone, clinical data such as symptoms and laboratory values are to be correlated with the image data and utilized by the algorithm. Among other things, this should increase the sensitivity, accuracy and specificity of image-based diagnostics in order to enable faster, non-invasive diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* Patients of any age or gender.
* CT scans confirming the presence of a retroperitoneal mass.
* Confirmed diagnosis of retroperitoneal fibrosis, sarcoma or other malignancies (i.e. lymphoma, germ cell tumors, metastasis, infections, ganglioneuromas) through pathology reports or clinical follow-up.

Exclusion Criteria:

* Poor quality CT scans where the region of interest is not clearly visible.
* Previous treatments or surgeries that might alter the radiomic features of the tumors.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients with retroperitoneal fibrosis, sarcoma or other retroperitoneal diseases who have pre-op abdominal ct scans of good quality.
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2023-11-01 (Actual); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Radiomic accuracy for retroperitoneal fibrosis | 6 months
  Accuracy of the algorithm in differentiating between retroperitoneal fibrosis and other retroperitoneal diseases

SECONDARY OUTCOMES:
Radiomic accuracy for retroperitoneal sarcomas | 10 Months
  Accuracy of the algorithm in differentiating between retroperitoneal sarcoma and other retroperitoneal diseases using CT images

CONTACTS AND LOCATIONS:
Locations (2):
- Peking University International Hospital, Beijing, China
- Universitätsklinikum Mannheim, Mannheim, Baden-Wurttemberg, Germany

IPD SHARING:
Plan to Share IPD: No